CLINICAL TRIAL: NCT02339831
Title: A Prospective, Randomized, Controlled, Single Center Study Evaluating the Clinical Performance of CAMOPED Following Knee Replacement
Brief Title: Active Versus Passive Motion Device Following Knee Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: The New England Baptist Hospital (Other)
Responsible Party: Principal Investigator, Wolfgang Fitz, Associate Orthopaedic Surgeon, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WFCAMCPM1
Record Dates: First submitted 2015-01-09; First posted 2015-01-16 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Knee Arthroplasty
Keywords: Knee; Arthroplasty; CPM; Camoped; Active vs Passive Motion Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- active motion device (Active Comparator): An active motion device (CAM) known as a CAMOPED was given after surgery. The device was used for 3 sessions of 20 minutes for 3 weeks.
  Interventions: Device: CAMOPED
- CPM passive motion device (Active Comparator): A continuous passive motion device (CPM) given after surgery. The device bends and moved the knee passively. It was used for 4 hours daily for 3 weeks.
  Interventions: Device: CPM passive motion device

INTERVENTIONS:
Device: CAMOPED — Camoped given after surgery
  Arms: active motion device
Device: CPM passive motion device — passive motion device given after surgery
  Arms: CPM passive motion device

SUMMARY:
The purpose of this study is to determine how well an active motion device, Camoped, works compared to a continuous passive motion device, CPM, for rehabilitation after partial or total knee replacement. It is hypothesized that the Camoped active motion device will provide outcomes equal to or superior than the CPM. Patients undergoing either partial or total knee replacement will be given the opportunity to participate. If they elect to participate, preoperative data will be collected including demographics, measures of strength, balance and knee bending, as well as surveys regarding current physical and mental health, as well as knee function. After surgery, patients will be randomly selected to receive either the Camoped or the CPM for use during their rehabilitation. After discharge, participants will be asked to maintain a daily diary tracking their use of the assigned device, as well as their daily pain levels. At a visit 4 weeks after surgery, participants will be asked to complete a series of surveys pertaining to their health and knee function, as well as to perform tests of strength, balance and knee bending. These results will be used to determine if one device produces superior rehabilitation results following total or partial knee replacement surgery.

DETAILED DESCRIPTION:
The purpose of this study is to determine how well an active motion device, Camoped, works compared to a continuous passive motion device, CPM, for rehabilitation after partial or total knee replacement. It is hypothesized that the Camoped active motion device will provide outcomes equal to or superior than the CPM. 110 patients will be randomized during the course of the study. Participation lasts approximately 4 weeks. Data for patients who begin the trial, but choose to drop out or are lost to follow up will not be included in analysis.

Patients who have elected to undergo surgery with one of the PIs, either a total knee replacement with Dr. Richard Scott or a partial knee replacement with Dr. Wolfgang Fitz, will be informed about the study and offered participation if they meet eligibility criteria. The PI will obtain written consent in the office for those who choose to participate. For participants, demographic data including height, weight, BMI, age and sex will be collected. Additionally, sit-to-stand, knee flexion, proprioception, strength and balance testing will be performed in the office by a physical therapist. Participant responses to the SF-36 physical and mental health surveys, knee function score, KSS and WOMAC questionnaires will also be collected.

Patients will be randomized to receive either the Camoped or CPM device after surgery. Patients will receive the device and its protocol for usage in the hospital following surgery. They will use the device for the duration of their hospital stay, and then take the device home. At home, patients will be asked to keep a daily diary tracking device usage as well as daily pain and medication intake. These results will be compared as part of the study analysis.

When patients return for their follow-up appointment four weeks after surgery, demographic data including height, weight, BMI, age and sex will be collected. Additionally, sit-to-stand, knee flexion, proprioception, strength and balance testing will be performed in the office. Participant responses to the SF-36 physical and mental health surveys, knee function score, KSS and WOMAC questionnaires will also be collected. These measures will be compared to the preoperative results.

Two-sample t-tests will be used to analyze the similarity between the two treatment groups before the intervention and to assess any differences afterwards. The Wilcoxon-Mann Whitney test will be performed as a non-parametric alternative to t-testing for any data sets found to be non-normal.

Data collection and management will be the responsibility of the PIs. All adverse events will be reported as necessary.

ELIGIBILITY:
Inclusion Criteria:

* • At least 18 years of age

  * Undergoing unilateral knee replacement
  * If female, not pregnant
  * Agree to participate in the follow-up appointment
  * Understand and sign the informed consent form

Exclusion Criteria:

* Bilateral UKA or TKA planned
* Cannot use non-operated leg post-operatively to propel active motion splint, caused by neurological or muscular diseases such as complete or incomplete paralysis or other causes of weakness with an inability to bend or extend knee
* Loss of sensation of/in? operated or non-operated leg
* Received investigational articles <30 days prior to enrollment or was currently receiving investigational products or devices.
* Below or above knee amputations of non-operated leg
* Below knee amputation of operated side
* Chronic pain syndrome with inability to walk and/or use active or passive motion device post-operatively
* Patients taking chronic narcotics and/or are taking more than 10mg codeine per day, or any Hydrocodone, more than 200 mg of tramadol, or any other narcotics prescribed for moderate to severe pain
* Patients involved in pain clinics for chronic pain, or pain that is not related to the knee
* Diagnosis of knee disorder other than osteoarthritis, post-traumatic osteoarthritis, gout, pseudo gout
* Inability to walk due to disorders unrelated to the knee (e.g., hip disorders, spinal stenosis, paralysis, hemiparalysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Fitz, MD, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mizner RL, Petterson SC, Stevens JE, Vandenborne K, Snyder-Mackler L. Early quadriceps strength loss after total knee arthroplasty. The contributions of muscle atrophy and failure of voluntary muscle activation. J Bone Joint Surg Am. 2005 May;87(5):1047-53. doi: 10.2106/JBJS.D.01992. PMID 15866968
- [Background] Harvey LA, Brosseau L, Herbert RD. Continuous passive motion following total knee arthroplasty in people with arthritis. Cochrane Database Syst Rev. 2010 Mar 17;(3):CD004260. doi: 10.1002/14651858.CD004260.pub2. PMID 20238330
- [Background] Arnold BL, Schmitz RJ. Examination of balance measures produced by the biodex stability system. J Athl Train. 1998 Oct;33(4):323-7. PMID 16558529
- [Background] Gstoettner M, Raschner C, Dirnberger E, Leimser H, Krismer M. Preoperative proprioceptive training in patients with total knee arthroplasty. Knee. 2011 Aug;18(4):265-70. doi: 10.1016/j.knee.2010.05.012. Epub 2010 Aug 30. PMID 20801047
- [Background] Wada M, Kawahara H, Shimada S, Miyazaki T, Baba H. Joint proprioception before and after total knee arthroplasty. Clin Orthop Relat Res. 2002 Oct;(403):161-7. doi: 10.1097/00003086-200210000-00024. PMID 12360022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1153 patients electing to undergo unilateral partial or total knee replacement at the New England Baptist Hospital from 03/2007-12/2010 were screened for participation. Of these patients, 110 elected to participate in the study and were randomized into one of the two study groups.
Groups:
- Active Motion Device: Patients assigned to this group receive the active motion device (CAM, Camoped) after surgery.
- Passive Motion Device: Patients assigned to this group receive the continuous passive motion device (CPM) after surgery.
Period: Overall Study
Arm/Group | Active Motion Device | Passive Motion Device
Started | 58 | 52
Lost to Follow Up | 20 | 7
Completed | 38 | 45
Not Completed | 20 | 7

BASELINE CHARACTERISTICS:
Population: 137 patients agreed to participate, 27 did not meet the inclusion criteria and 110 signed the informed consent form. Following allocation to their group, we excluded 24 patients (20 using CAM and 7 CPM) who did not finish the study due to non-compliance, leaving a total of 83 patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Motion Device | Passive Motion Device | Total
Number analyzed (Participants) | 38 | 45 | 83
Age, Continuous [Median (Standard Deviation); unit: years] | 61.5 (8.8) | 64.7 (9.2) | 63.2 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 31 | 51
  Male | 18 | 14 | 32
Kinesthesia [Mean (Standard Deviation); unit: degrees] — Kinesthesia was measured by recording the angle of the flexed knee and documenting how close the patient was able to reproduce the angle with closed eyes. The differences were recorded in degrees using an 8-inch goniometer.
  degrees | 3.20 (2.64) | 4.24 (3.34) | 3.7 (3.0)
Quadriceps Strength [Mean (Standard Deviation); unit: newton meter] | 12.4 (4.7) | 11.2 (4.7) | 11.8 (4.7)
Balance [Mean (Standard Deviation); unit: units on a scale] — Biodex Balance Machine Score. The system consists of a multiaxial standing platform with a maximum tilt of 20 degrees. All participants were tested on level 8, and a balance index was calculated using the time and deviation (in degrees) on the platform relative to a neutral position. The normal range for adults 54-71 is 1.79 - 3.35. Lower values indicate better/greater stability.
  units on a scale | 3.61 (1.69) | 3.62 (1.39) | 3.62 (1.53)
Knee Flexion [Mean (Standard Deviation); unit: degrees] — Knee-flexion was measured using an 8-inch goniometer.
  degrees | 113.8 (12.8) | 111.6 (12.8) | 112.6 (12.8)
SF-36 Mental Health Score [Mean (Standard Deviation); unit: units on a scale] — Short form 36 mental health score. The scale is measured from 0-100. 0 is the lowest or worst possible level of functioning and 100 is the highest or best possible level of functioning.
  units on a scale | 43.4 (7.5) | 43.2 (8.1) | 43.3 (7.8)
Knee Society Score [Mean (Standard Deviation); unit: units on a scale] — Knee society score is an objective patient reported outcome survey to measure a patient's functional ability before and after knee arthroplasty. It is measured on a scale of 1-100. A score between 80-100 indicated excellent functioning, a score between 70-79 indicates good functioning, a score between 60-69 indicates fair functioning, and a score below 60 indicates poor functioning.
  units on a scale | 56.0 (13.7) | 49.3 (14.9) | 54.7 (17.8)
WOMAC [Mean (Standard Deviation); unit: units on a scale] — Western Ontario and McMaster Universities Arthritis Index is measured on a scale of 0-68. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
  units on a scale | 64.1 (14.9) | 67.1 (20.3) | 65.7 (17.7)
Sit-to-Stand Test [Mean (Standard Deviation); unit: seconds] — After one demonstration of the sit-to-stand test, standing up from a seated position without support, two tests were timed and the better value recorded.The patient was directed to sit with his/her back against the chair and arms crossed in front. Time started when timer said "Go".
  seconds | 3.37 (1.18) | 3.40 (1.48) | 3.39 (1.34)
SF-36 Physical Health Score [Mean (Standard Deviation); unit: units on a scale] — Short form 36 is a patient reported outcome survey used to asses physical health. The scale is 0-100. Lower scores indicate more disability and higher scores indicate less disability.
  units on a scale | 35.1 (6.3) | 35.0 (6.8) | 35.0 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Early Functional Outcome Strength
Description: Quadriceps strength measurements using a hand held dynamometer
Time Frame: 4-6 weeks post-op
Measure: Mean (Standard Deviation); unit: newton meter
Arm/Group | Active Motion Device | Passive Motion Device
Number analyzed (Participants) | 38 | 45
newton meter | 12.02 (4.12) | 11.60 (4.34)

2. Primary Outcome: Early Functional Outcome by Sit to Stand Test
Description: Sit-to-Stand test: After one demonstration of the sit-to-stand test, standing up from a seated position without support, two tests were timed and the better value recorded. Patient was asked to sit with back against chair and told to stand up without using any support. Arms were suggested to be folded in front of chest. Time started with recorded said "Go".
Time Frame: 4-6 weeks post-op
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active Motion Device | Passive Motion Device
Number analyzed (Participants) | 38 | 45
seconds | 2.83 (.98) | 3.43 (1.23)

3. Primary Outcome: Early Functional Outcome Proprioception
Description: Biodex Balance Machine Score. The system consists of a multiaxial standing platform with a maximum tilt of 20 degrees. All participants were tested on level 8, and a balance index was calculated using the time and deviation (in degrees) on the platform relative to a neutral position. The normal range for adults 54-71 is 1.79 - 3.35. Lower values indicate better/greater stability.
Time Frame: 4-6 weeks post-op
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Motion Device | Passive Motion Device
Number analyzed (Participants) | 38 | 45
units on a scale | 3.11 (1.56) | 2.98 (1.27)

4. Primary Outcome: Early Function Outcome Kinesthesia
Description: Kinesthesia was measured by recording the angle of the flexed knee and documenting how close the patient was able to reproduce the angle with closed eyes. The differences were recorded in degrees using an 8-inch goniometer.
Time Frame: 4-6 weeks post op
Measure: Mean (Standard Deviation); unit: degress
Arm/Group | Active Motion Device | Passive Motion Device
Number analyzed (Participants) | 38 | 45
degress | 2.90 (2.99) | 2.98 (2.32)

5. Primary Outcome: Early Functional Outcome Knee Flexion
Description: Knee-flexion was measured using an 8-inch goniometer.
Time Frame: 4-6 weeks post op
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Active Motion Device | Passive Motion Device
Number analyzed (Participants) | 38 | 45
degrees | 104.3 (15.0) | 101.0 (12.7)

6. Secondary Outcome: General Mental Orthopaedic Outcome Measures
Description: Short form 36 mental health score. The scale is measured from 0-100. 0 is the lowest or worst possible level of functioning and 100 is the highest or best possible level of functioning.
Time Frame: 4-6 weeks post-op
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Motion Device | Passive Motion Device
Number analyzed (Participants) | 38 | 45
units on a scale | 40.2 (8.8) | 39.4 (8.2)

7. Secondary Outcome: General Activity Orthopaedic Outcome Measures
Description: Western Ontario and McMaster Universities Arthritis Index is measured on a scale of 0-68. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Time Frame: 4-6 weeks post-op
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Motion Device | Passive Motion Device
Number analyzed (Participants) | 38 | 45
units on a scale | 45.8 (13.6) | 50.2 (16.9)

8. Secondary Outcome: General Functional Orthopaedic Outcome Measures
Description: Knee society score is an objective patient reported outcome survey to measure a patient's functional ability before and after knee arthroplasty. It is measured on a scale of 1-100. A score between 80-100 indicated excellent functioning, a score between 70-79 indicates good functioning, a score between 60-69 indicates fair functioning, and a score below 60 indicates poor functioning.
Time Frame: 4-6 weeks post-op
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Motion Device | Passive Motion Device
Number analyzed (Participants) | 38 | 45
units on a scale | 64.7 (17.0) | 62.6 (17.7)

9. Secondary Outcome: General Pain
Description: Self-reported total pain medication consumption was recorded by patients and at the end of the four-week period converted into standard units for comparison as "oxycodone equivalent dosage".
Time Frame: 4-6 weeks post-op
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Motion Device | Passive Motion Device
Number analyzed (Participants) | 38 | 45
mg | 471.77 (457.46) | 346.97 (289.85)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected while patients were participating the study. Patients were followed up at 4 weeks after surgery and any adverse events were noted.
Arm/Group | Active Motion Device | Passive Motion Device
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/45
Other Adverse Events (participants affected / at risk) | 0/38 | 0/45

LIMITATIONS AND CAVEATS:
We ran into an unexpected problem in recruiting patients for this study. Many did not want to participate in this study, as they did not want to use the passive device and were not willing to use it 4 hours each day.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No